CLINICAL TRIAL: NCT04259593
Title: Exercise Training is a Feasible and Active Complementary Therapy in Adult and Elderly Patients Receiving Anti- Lymphoma Treatments
Brief Title: Exercise for Elderly Lymphoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mario Vetrano, MD, MD, PhD, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 553
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Elderly Lymphoma Patients
Keywords: Exercise training, Complementary therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training Group (Experimental): Exercise training group performed three weekly sessions for 16 weeks. This program consisted of moderate intensity aerobic, resistance, balance, and stretching exercises. The duration of every exercise session was 35 minutes during the first week and 65 minutes from the second week onward.
  Interventions: Other: exercise training
- Control Group (No Intervention): The control group received usual lymphoma care

INTERVENTIONS:
Other: exercise training
  Arms: Exercise Training Group

SUMMARY:
This pilot study was designed in a real-life setting to establish the feasibility, the safety and the activity of a supervised and combined Exercise Training (ET) program in adult and elderly lymphoma patients undergoing cancer-treatments.

DETAILED DESCRIPTION:
Eligible patients were assigned to the ET group. All the patients eligible for exercise but not partiticpating to the ET program because of logistical reasons, were considered as the control group. All clinical outcomes were assessed before exercise training (T0), 3 (T1) and 6-months (T2) after the beginning of the exercise.

ELIGIBILITY:
Inclusion Criteria:

* ≥18-80 years old, histologically conﬁrmed HL or NHL, patients in need of first or subsequent lines of systemic treatment and with a long-life expectancy

Exclusion Criteria:

* Patients were excluded if they had less than 4 months of anti-cancer treatment to be delivered, severe orthopaedic, cardiac, pulmonary, or cognitive impairment, osteolytic lesions with the risk of fracture, cachexia or if they were ≥ 65 years and frail on the basis of comprehensive geriatric assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
The eligibility rate | 6 months
  the eligibility rate was assessed by the number of eligible patients divided by the total number of elements on the sampling frame.
The recruitment rate | 6 months
  the recruitment rate was assessed by the number of patients included in the study divided by the total number of eligible patients
The exercise adherence rate | 4 months
  The exercise adherence rate was assessed by the number of exercise sessions attended out of the 48 sessions scheduled for each patient
The assessment rate | 6 months
  The assessment rate was assessed by the number of patients who completed the T1 and T2 follow-up times over the total number who participated in the study
Safety of the exercise training | 6 months
  Safety was assessed by monitoring any serious adverse events that occured during the ET period.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Christina Cox, Study Chair — Sant'Andrea Hospital, Rome, Italy
Locations (1):
- Sant'Andrea Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Streckmann F, Kneis S, Leifert JA, Baumann FT, Kleber M, Ihorst G, Herich L, Grussinger V, Gollhofer A, Bertz H. Exercise program improves therapy-related side-effects and quality of life in lymphoma patients undergoing therapy. Ann Oncol. 2014 Feb;25(2):493-9. doi: 10.1093/annonc/mdt568. PMID 24478323